CLINICAL TRIAL: NCT03170193
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Ascending Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 529 in Healthy Subjects
Brief Title: AMG 529 First in Human Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20160338
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular

STUDY DESIGN:
Intervention Model Description: Within each dose cohort participants were randomized in a 3:1 ratio to receive either AMG 529 or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMG 529 (Experimental): Participants received a single dose of AMG 529 at ascending dose levels by either subcutaneous or intravenous injection.
  Interventions: Drug: AMG 529
- Placebo (Placebo Comparator): Participants received a single dose of placebo matching to AMG 529 by either subcutaneous or intravenous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 529 — Ascending single doses of AMG 529 by subcutaneous (SC) or intravenous (IV) injection
  Arms: AMG 529
Drug: Placebo — Single doses of matching placebo by SC or IV injection
  Arms: Placebo

SUMMARY:
A study to assess the safety and tolerability of AMG 529 following single, ascending doses administered subcutaneously (SC) or intravenously (IV) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women ≥ 18 to ≤ 55 years old with no history or evidence of clinically relevant medical disorders
2. Body mass index (BMI) between 18 and 32 kg/m², inclusive, at screening
3. Women must be of non-reproductive potential as defined in protocol
4. Other inclusion criteria may apply

Exclusion Criteria:

1. Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives (whichever is longer), since ending treatment on another investigational device or drug study(s) prior to receiving the first dose of investigational product
2. Women who are lactating/breastfeeding or who plan to breastfeed while on study through 90 days after receiving the dose of investigational product
3. Men with partners who are pregnant or planning to become pregnant while the subject is on study through 90 days after receiving the dose of investigational product
4. Positive pregnancy test at screening or day -1
5. Other exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States. Participants were enrolled from 15 May 2017 to 18 September 2017.
Pre-assignment Details: Participants were enrolled into one of six dose cohorts. Within each cohort participants were randomized in a ratio of 3:1 to receive AMG 529 or placebo.
Groups:
- Placebo: Participants received a single dose of matching placebo by either subcutaneous or intravenous injection.
- AMG 529 21 mg SC: Participants received a single dose of 21 mg AMG 529 on study day 1 by subcutaneous (SC) injection.
- AMG 529 70 mg SC: Participants received a single dose of 70 mg AMG 529 on study day 1 by subcutaneous injection.
- AMG 529 210 mg SC: Participants received a single dose of 210 mg AMG 529 on study day 1 by subcutaneous injection.
- AMG 529 420 mg SC: Participants received a single dose of 420 mg AMG 529 on study day 1 by subcutaneous injection.
- AMG 529 700 mg SC: Participants received a single dose of 700 mg AMG 529 on study day 1 by subcutaneous injection.
- AMG 529 70 mg IV: Participants received a single dose of 70 mg AMG 529 on study day 1 by intravenous (IV) injection.
Period: Overall Study
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 11 | 5 | 6 | 5 | 6 | 6 | 6
Not Completed | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.5) | 33.5 (12.5) | 32.3 (11.6) | 45.2 (11.6) | 35.0 (11.0) | 36.5 (9.6) | 34.7 (12.7) | 36.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Male | 12 | 6 | 6 | 5 | 6 | 6 | 5 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 6
  Not Hispanic or Latino | 9 | 5 | 5 | 6 | 6 | 5 | 6 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 5 | 5 | 5 | 2 | 3 | 4 | 5 | 29
  White | 7 | 1 | 1 | 4 | 3 | 2 | 1 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Determination of the severity of adverse events was according to the following: grade 1 = mild (eg, asymptomatic or mild symptoms); grade 2 = moderate (eg, minimal intervention indicated or interferes with activity); grade 3 = severe (eg, medically significant but not immediately life-threatening, prevents daily activity, or requires treatment); grade 4 = life-threatening (ie, refers to an event in which the participant was, in the view of the investigator, at risk of death at the time of the event); and grade 5 = fatal.
  A serious adverse event was defined as an adverse event that met at least 1 of the following criteria:
  * fatal
  * life threatening
  * required in patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event.
Time Frame: From first dose up to 30 days for participants assigned to the 21 mg or 70 mg dose cohorts and up to 57 days for participants assigned to the 210 mg, 420 mg, or 700 mg dose cohorts.
Population: Randomized participants who received at least 1 dose of AMG 529 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  All adverse events | 3 | 0 | 0 | 2 | 2 | 3 | 2
  Adverse events Grade ≥ 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Adverse events Grade ≥ 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adverse events Grade ≥ 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse events | 1 | 0 | 0 | 2 | 2 | 0 | 2
  Fatal adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 529
Time Frame: Predose and at 0.5 and 1 hour postdose (IV cohort only) and 6, 12, 24, 36, 48, 72, 120, 168, 240, 366, 504, and 696 hours postdose (all participants) and additionally at days 43 and 57 for participants assigned to the 210, 420, or 700 mg dose cohorts.
Population: Participants who received AMG 529 for whom at least 1 PK parameter or endpoint was reliably estimated. Four participants were excluded from PK analyses as their profiles had < 2 samples that were above the lower limit of quantification.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6 | 6
ng/mL | 6.90 (1.73) | 23.8 (13.4) | 2010 (3120) | 9370 (10800) | 35600 (32700) | 3460 (4430)

3. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of AMG 529
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6 | 6
hours | 24 [12 to 24] | 5.8 [5.8 to 5.8] | 72 [24 to 72] | 72 [24 to 72] | 96 [36 to 170] | 0.5 [0.5 to 0.5]

4. Secondary Outcome: Area Under the Curve From Time 0 to the Last Quantifiable Concentration (AUClast) for AMG 529
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days*ng/mL
Arm/Group | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6 | 6
days*ng/mL | 5.99 (2.90) | 46.0 (47.4) | 5370 (8520) | 41800 (51000) | 289000 (330000) | 766 (1240)

5. Secondary Outcome: Change From Baseline in Blood Alkaline Phosphatase Concentration Over Time
Time Frame: Baseline and days 3, 8, and 30
Population: Participants who received at least 1 dose of study drug and with available data at each time point
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
units/liter
  Baseline | 62.0 (13.8) | 69.0 (21.2) | 56.0 (10.8) | 68.0 (12.2) | 57.7 (9.0) | 57.5 (18.0) | 58.0 (8.1)
  Change from baseline to day 3 | -0.3 (4.2) | 4.7 (4.7) | 7.0 (7.0) | 57.0 (51.7) | 76.7 (76.9) | 88.2 (33.5) | 28.7 (14.7)
  Change from baseline to day 8: number analyzed (Participants) | 12 | 6 | 6 | 5 | 6 | 6 | 5
  Change from baseline to day 8 | 2.3 (6.0) | 3.2 (7.5) | 17.0 (10.4) | 102.6 (70.8) | 199.3 (256.1) | 155.8 (34.8) | 8.8 (5.8)
  Change from baseline to day 30: number analyzed (Participants) | 11 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 30 | 3.5 (8.5) | -1.4 (4.0) | 1.8 (5.3) | -0.8 (4.0) | 11.8 (5.9) | 14.6 (6.5) | 2.0 (7.8)

6. Secondary Outcome: Change From Baseline in Total Cholesterol Concentration Over Time
Time Frame: Baseline and days 3, 6, 11, 22, 30 (all participants), and day 57 for participants assigned to the 210 mg, 420 mg, or 700 mg cohorts.
Population: Randomized participants who received study drug with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
mmol/L
  Baseline | 4.5817 (0.8204) | 5.3567 (0.9662) | 4.8383 (1.0789) | 5.3417 (0.9771) | 4.2483 (0.6335) | 4.8533 (0.8125) | 5.0633 (1.5937)
  Change from baseline to day 3 | 0.0692 (0.2381) | -0.1583 (0.1347) | -0.0200 (0.2254) | 0.0800 (0.2224) | 0.1617 (0.2375) | 0.2350 (0.1299) | 0.3400 (0.3428)
  Change from baseline to day 6: number analyzed (Participants) | 12 | 6 | 6 | 5 | 6 | 6 | 6
  Change from baseline to day 6 | 0.0867 (0.4151) | -0.3317 (0.1997) | -0.3533 (0.3426) | -0.2520 (0.6208) | -0.3267 (0.3140) | -0.1667 (0.2614) | 0.3350 (0.5461)
  Change from baseline to day 11: number analyzed (Participants) | 12 | 5 | 6 | 5 | 6 | 4 | 5
  Change from baseline to day 11 | -0.4625 (0.4110) | -1.0620 (0.5976) | -0.6933 (0.4763) | -0.6700 (0.5770) | -0.8500 (0.6339) | -0.7600 (0.5306) | -0.0340 (0.8344)
  Change from baseline to day 22: number analyzed (Participants) | 12 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 22 | -0.0300 (0.5567) | -0.7480 (0.8825) | -0.2550 (0.5021) | -0.1640 (0.3092) | -0.2183 (0.4100) | -0.2040 (0.5358) | -0.3200 (0.9193)
  Change from baseline to day 30: number analyzed (Participants) | 11 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 30 | -0.0936 (0.7880) | -0.6780 (0.3467) | -0.1933 (0.4376) | 0.1300 (0.0919) | 0.2583 (0.4088) | 0.1380 (0.4964) | -0.1140 (0.9209)
  Change from baseline to day 57: number analyzed (Participants) | 5 | 0 | 0 | 5 | 6 | 6 | 0
  Change from baseline to day 57 | 0.1840 (0.7451) |  |  | 0.5120 (0.8889) | 0.2383 (0.4896) | -0.0033 (0.9705) |

7. Secondary Outcome: Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) Concentration Over Time
Time Frame: as for outcome 6
Population: Randomized participants who received study drug with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
mmol/L
  Baseline | 2.8317 (0.8071) | 3.2683 (1.0026) | 2.8400 (0.7687) | 3.4017 (1.2875) | 2.4633 (0.5727) | 3.2267 (0.7112) | 3.1583 (1.1382)
  Change from baseline to day 3 | 0.1608 (0.2423) | 0.1383 (0.3271) | 0.2150 (0.1571) | -0.0867 (0.3280) | 0.2650 (0.1401) | 0.3350 (0.2482) | 0.3350 (0.2874)
  Change from baseline to day 6: number analyzed (Participants) | 12 | 6 | 6 | 5 | 6 | 6 | 6
  Change from baseline to day 6 | 0.1400 (0.2992) | 0.0417 (0.3547) | 0.1050 (0.1549) | -0.5860 (0.5180) | -0.0967 (0.2708) | -0.0967 (0.1975) | 0.1650 (0.5853)
  Change from baseline to day 11: number analyzed (Participants) | 12 | 5 | 6 | 5 | 6 | 4 | 5
  Change from baseline to day 11 | -0.3367 (0.4298) | -0.7600 (0.4464) | -0.3900 (0.2912) | -0.7920 (0.4873) | -0.7333 (0.5000) | -0.5850 (0.2204) | -0.0520 (0.5955)
  Change from baseline to day 22: number analyzed (Participants) | 12 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 22 | 0.0117 (0.4577) | -0.5240 (0.8043) | -0.0600 (0.3205) | -0.2860 (0.4116) | -0.3517 (0.3969) | -0.3960 (0.1521) | -0.2780 (0.7706)
  Change from baseline to day 30: number analyzed (Participants) | 11 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 30 | -0.1018 (0.6698) | -0.4260 (0.4258) | -0.0767 (0.4002) | -0.4020 (0.4773) | 0.2667 (0.3768) | -0.0740 (0.4999) | -0.2680 (0.9091)
  Change from baseline to day 57: number analyzed (Participants) | 5 | 0 | 0 | 5 | 6 | 6 | 0
  Change from baseline to day 57 | 0.0500 (0.7559) |  |  | 0.0520 (0.6514) | 0.1283 (0.3075) | -0.1617 (0.8583) |

8. Secondary Outcome: Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) Concentration Over Time
Time Frame: as for outcome 6
Population: Randomized participants who received study drug with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
mmol/L
  Baseline | 1.1775 (0.2932) | 1.3783 (0.2928) | 1.3950 (0.2626) | 1.4133 (0.4968) | 1.2633 (0.2202) | 1.0700 (0.4527) | 1.4417 (0.5517)
  Change from baseline to day 3 | -0.0592 (0.1094) | -0.0100 (0.1092) | -0.1267 (0.0935) | 0.0417 (0.1032) | -0.0600 (0.1373) | 0.0783 (0.0981) | -0.0383 (0.1118)
  Change from baseline to day 6: number analyzed (Participants) | 12 | 6 | 6 | 5 | 6 | 6 | 6
  Change from baseline to day 6 | -0.0975 (0.1096) | -0.1617 (0.1254) | -0.2083 (0.1430) | -0.0980 (0.1417) | -0.1100 (0.2028) | 0.0350 (0.1816) | -0.0767 (0.1402)
  Change from baseline to day 11: number analyzed (Participants) | 12 | 5 | 6 | 5 | 6 | 4 | 5
  Change from baseline to day 11 | -0.0133 (0.1224) | -0.2080 (0.1854) | -0.1600 (0.1689) | -0.0960 (0.1318) | -0.0800 (0.0812) | 0.0475 (0.0768) | -0.0060 (0.1809)
  Change from baseline to day 22: number analyzed (Participants) | 12 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 22 | 0.0208 (0.1468) | -0.0580 (0.1644) | -0.0417 (0.1815) | 0.0220 (0.1026) | 0.0583 (0.1533) | 0.2860 (0.1704) | 0.0320 (0.1583)
  Change from baseline to day 30: number analyzed (Participants) | 11 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 30 | 0.0473 (0.1769) | -0.0760 (0.0853) | -0.0400 (0.3107) | 0.1380 (0.1644) | 0.0667 (0.2060) | 0.2480 (0.0944) | 0.1340 (0.1396)
  Change from baseline to day 57: number analyzed (Participants) | 5 | 0 | 0 | 5 | 6 | 6 | 0
  Change from baseline to day 57 | -0.0540 (0.1549) |  |  | 0.1160 (0.1595) | 0.1483 (0.1113) | 0.2633 (0.2470) |

9. Secondary Outcome: Change From Baseline in Triglycerides Concentration Over Time
Time Frame: as for outcome 6
Population: Randomized participants who received study drug with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
mmol/L
  Baseline | 1.2292 (0.5080) | 1.1100 (0.5588) | 1.0050 (0.5478) | 1.3750 (0.9770) | 1.0533 (0.3525) | 1.5067 (1.0848) | 0.8317 (0.3036)
  Change from baseline to day 3 | -0.0942 (0.2880) | -0.1283 (0.1379) | -0.0633 (0.2366) | -0.0183 (0.3725) | -0.1833 (0.0993) | -0.5600 (0.6615) | 0.0750 (0.1244)
  Change from baseline to day 6: number analyzed (Participants) | 12 | 6 | 6 | 5 | 6 | 6 | 6
  Change from baseline to day 6 | -0.0525 (0.3015) | -0.0450 (0.1148) | -0.0583 (0.1932) | 0.4580 (1.2469) | -0.2900 (0.2521) | -0.5783 (0.5958) | 0.3133 (0.3102)
  Change from baseline to day 11: number analyzed (Participants) | 12 | 5 | 6 | 5 | 6 | 4 | 5
  Change from baseline to day 11 | -0.0975 (0.3470) | 0.2040 (0.7577) | 0.1400 (0.4963) | 0.1840 (0.4797) | -0.1167 (0.4131) | -0.5925 (1.0357) | 0.3320 (0.5496)
  Change from baseline to day 22: number analyzed (Participants) | 12 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 22 | 0.0475 (0.5965) | 0.0920 (0.2212) | 0.5800 (0.6549) | 0.1780 (0.4043) | 0.2183 (0.2193) | -0.4360 (0.9239) | 0.3340 (0.4185)
  Change from baseline to day 30: number analyzed (Participants) | 11 | 5 | 6 | 5 | 6 | 5 | 5
  Change from baseline to day 30 | 0.0991 (0.4538) | 0.2320 (0.3214) | 0.5533 (0.7672) | 0.2600 (0.5742) | 0.0533 (0.4320) | -0.0360 (0.5330) | 0.2220 (0.1580)
  Change from baseline to day 57: number analyzed (Participants) | 5 | 0 | 0 | 5 | 6 | 6 | 0
  Change from baseline to day 57 | 0.4580 (0.5334) |  |  | 0.4900 (0.7883) | 0.0533 (0.3663) | -0.3283 (0.5669) |

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days for participants assigned to the 21 mg or 70 mg dose cohorts and up to 57 days for participants assigned to the 210 mg, 420 mg, or 700 mg dose cohorts.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | AMG 529 21 mg SC | AMG 529 70 mg SC | AMG 529 210 mg SC | AMG 529 420 mg SC | AMG 529 700 mg SC | AMG 529 70 mg IV
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/12 | 0/6 | 0/6 | 2/6 | 2/6 | 3/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | AMG 529 21 mg SC (N=6) | AMG 529 70 mg SC (N=6) | AMG 529 210 mg SC (N=6) | AMG 529 420 mg SC (N=6) | AMG 529 700 mg SC (N=6) | AMG 529 70 mg IV (N=6)
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03170193/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT03170193/SAP_001.pdf